CLINICAL TRIAL: NCT00227474
Title: S0348: A Phase II Study of 5T4-Modified Vaccinia Ankara (MVA) Vaccine (TROVAX) in Patients With Advanced Breast Cancer
Brief Title: S0348 Vaccine Therapy in Treating Patients With Stage IIIB or Stage IV Breast Cancer in Remission
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: SWOG has decided to not pursue this trial
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441167; S0348 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: recombinant modified vaccinia Ankara-5T4 vaccine
Procedure: adjuvant therapy
Procedure: recombinant viral vaccine therapy

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells. Giving booster vaccinations may make a stronger immune response and prevent or delay the recurrence of cancer.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with stage IIIB or stage IV breast cancer in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of conducting a live viral vaccine trial using adjuvant recombinant modified vaccinia Ankara-5T4 vaccine (TroVax®) in patients with stage IIIB-IV breast cancer in remission.
* Determine the progression-free survival of patients treated with this vaccine.
* Determine the 5T4-specific T-cell immune response in patients treated with this vaccine.
* Determine the toxicity of this vaccine in these patients.
* Determine the level of 5T4-specific antibody response in patients treated with this vaccine.
* Correlate, preliminarily, immune response with 3- and 12-month progression-free survival of patients treated with this vaccine.
* Correlate tumor 5T4 expression with overall survival and progression-free survival of patients treated with this vaccine.
* Correlate tumor infiltrating lymphocyte and CD1a-positive dendritic cell density with development of 5T4-specific T-cell immunity in patients treated with this vaccine.

OUTLINE: This is a multicenter study.

Patients receive recombinant modified vaccinia Ankara-5T4 vaccine (TroVax®) intramuscularly once a month in months 1-3. Patients then receive booster vaccinations once in months 6, 9, and 12. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage IIIB-IV disease

    * Patients with stage IV disease must have metastasis to the bone only AND documentation of negative or improved bone scan showing evidence of recalcification by plain film x-ray OR MRI showing normalization of marrow signal
* In remission (no evidence of disease)

  * Must have completed appropriate treatment (e.g., radiotherapy and chemotherapy) for primary disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No known history of hepatitis B or C

Renal

* Not specified

Immunologic

* No known HIV positivity
* No known history of immune-deficiency disorder
* No history of allergic reaction to prior vaccinia vaccinations
* No autoimmune disease requiring concurrent treatment

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Concurrent trastuzumab (Herceptin®) allowed provided it is not part of treatment on another clinical trial

Chemotherapy

* See Disease Characteristics
* At least 28 days since prior cytotoxic chemotherapy

Endocrine therapy

* At least 28 days since prior steroid therapy
* Concurrent hormonal therapy allowed provided it is not part of treatment on another clinical trial

Radiotherapy

* See Disease Characteristics
* At least 28 days since prior radiotherapy

Surgery

* Not specified

Other

* At least 28 days since prior and no concurrent treatment on another clinical trial

  * Patients enrolled in a SWOG phase III metastatic trial (e.g.,SWOG-S0226 or SWOG-S0347) who have achieved complete remission but not yet progressed are not eligible
  * Patients enrolled in a SWOG phase II metastatic trial or phase II/III adjuvant or neoadjuvant trial (e.g., SWOG-S0012, SWOG-S0215, SWOG-S0221, SWOG-S0338, or SWOG-S0430) who have achieved complete remission/no evidence of disease status and are no longer receiving study treatment are eligible
* Concurrent bisphosphonates allowed provided it is not part of treatment on another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lupe G. Salazar, MD, Study Chair — Tumor Vaccine Group at the University of Washington; Mary (Nora) L. Disis, MD, Study Chair — University of Washington